CLINICAL TRIAL: NCT05496010
Title: Comparing the Effectiveness of Dry Needling and Ischemic Compression Technique on Muscle Thickness and Health Related Quality of Life in Trigger Point Tension Type Headache
Brief Title: Comparing the Effectiveness of Dry Needling and Ischemic Compression on Tension Type Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Aribah Ahmed, MPhil Candidate ZCRS, Ziauddin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4541121AAREH
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Tension-Type Headache
MeSH Terms: conditions — Tension-Type Headache | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: Group A: Dry Needling treatment given for 6 sessions, 3 days/week for 2 weeks on the trigger points located in Upper Trapezius, Sternocleidomastoid, Sub occipitalis and Temporalis muscles.
  Group B:
  Ischemic Compression technique given for 6 sessions, 3 days/week for 2 weeks on the trigger points located in Upper Trapezius, Sternocleidomastoid, Sub occipitalis and Temporalis muscles.
Who Masked: Participant
Masking Description: All participants will be blinded regarding treatment. A total of 30 patients will be recruited and assigned into two groups. Group A will receive Dry needling sessions and group B will receive Ischemic compression technique.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling (Experimental): Dry needling will be performed on the patients of group A after the diagnosis of trigger points in particular muscles.The complete treatment session will be comprised of 3 sessions per week for two weeks followed by follow up after 1 month until the symptoms have been improved.
  Interventions: Other: Dry Needling and Ischemic Compression Technique
- Ischemic Compression Technique (Active Comparator): Ischemic Compression technique will be performed on the patients of group B after the diagnosis of trigger points in particular muscles by diagnostic ultrasound. The complete treatment session will be comprised of 3 sessions per week for two weeks followed by follow up after 1 month until the symptoms have been improved.
  Interventions: Other: Dry Needling and Ischemic Compression Technique

INTERVENTIONS:
Other: Dry Needling and Ischemic Compression Technique — For Group A, Dry needling will be applied into trigger points which are active and present in the muscles, efficiently and within the safe limits taking all the safety precautions.
  For group B, Ischemic Compression Technique will be applied on trigger points.
  The complete treatment session will be comprised of 3 sessions per week for two weeks followed by follow up after 1 month until the symptoms have been improved for both the groups.

SUMMARY:
Headaches are the main health problem as one of the prevalent type of all symptoms in the world population. Among different types of headaches, the most prevailing primary headache in general population is Tension-type headache (TTH). According to Global Burden Disease study conducted in 2016 tension-type headache ranks the third highest primary headache syndromes among 32 diseases and injuries in 195 countries from the Period of 1990 to 2016.These types of headaches are associated with significant reductions in productivity of an individual with prominent increase in socioeconomic costs. There are various treatments suggested for improving the symptoms in trigger point related tension type headaches such as usage of hot packs, cryotherapy, ultrasound therapy, mobilization and manipulation techniques, Dry needling, MET and ICT. None of the study has been conducted in Pakistan which has compared two specific techniques to resolve trigger points with the accuracy of diagnosis by diagnostic ultrasound in limited time period, which is cost friendly, and provides quick relief to patients without causing a lot of pain. Therefore, more studies are needed to overcome the gap area in the use of specific techniques in clinics with accurate diagnosis by the clinicians of Pakistan.

DETAILED DESCRIPTION:
The research aims to compare the effectiveness of Dry Needling and Ischemic Compression Technique on muscle thickness & health related quality of life in trigger point related tension type headache. Headaches are the major health concern as one of the prevalent type of all symptoms in the worldwide population and are the cause of disabilities and hindrance in productivity of an individual.

The treatment approaches performed for trigger point related tension type headache are non-specific, vigorous, time consuming and costly. It is due to the inaccurate location of the trigger points present in cervical musculature. The studies related to comparison of specific treatment procedures to treat trigger point related tension type headaches such as dry needling and Ischemic Compression technique with the knowledge of accurate location of trigger points present in cervical musculature are lacking in Pakistani population. Hence the current study is aimed to determine the effect of dry needling and Ischemic Compression technique with the use of diagnostic ultrasound on muscle thickness, pain and health related quality of life in Trigger point related tension type headache. The study will be conducted on the tension type headache diagnosed individuals aged 20 to 50 years of age, at Physical Therapy OPD of Saifee and Ziauddin Hospital with the help of envelope method as a randomization technique. Dry needling will be performed on Group A whereas Group B will be given Ischemic Compression technique on trigger points diagnosed by Musculoskeletal Ultrasound. Patient's headache, muscle thickness and health related quality of life will be assessed by Numeric Pain rating scale, Musculoskeletal Ultrasound and Short Form-36 Questionnaire respectively. If the data will be found to be normally distributed, Pair T-test will be run for with the group analysis. Between the groups an alysis will be perform by Independent t test. In case data found to be deviated from the assumption of normal distribution, Paired T-test will be replaced by Wilcoxon test and Independent T test will be replaced by Mann Whitney U Test. The level of significance will be kept at 95% alpha-0.05.

ELIGIBILITY:
Inclusion Criteria:

* 20-50 aged individuals years
* Trigger point related Tension Type Headache diagnosed by Neurologist.
* Patients having trigger points in the muscles taken in the study.

Exclusion Criteria:

* Medical Red flags
* Major Depression
* Neurological or Cardiovascular Disease.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale to assess headache intensity | Baseline
  Pain will be assessed through Numeric Pain Rating Scale NPRS among trigger point tension type headache individuals, where high values indicate greater pain intensity.
Numeric Pain Rating Scale to assess headache intensity | After 2 weeks
  Pain will be assessed through Numeric Pain Rating Scale NPRS among trigger point tension type headache individuals where high values indicate greater pain intensity.
Short Form-36 Questionnaire to measure Health related quality of life. | Pre-Treatment
  All the domains of Health related quality of life assessment will be carried out through the individual's scoring.
Short Form-36 Questionnaire to measure Health related quality of life | After 2 weeks. (Follow up)
  All the domains of Health related quality of life assessment will be carried out through the individual's scoring.
Diagnostic Ultrasound to measure muscle thickness | Pre-Treatment
  An ultrasound examination will be performed to find out the muscle thickness of cervical muscles in which trigger points are present.
Diagnostic Ultrasound to measure muscle thickness | After 2 weeks. (Follow up)
  An ultrasound examination will be performed to find out the muscle thickness of cervical muscles in which trigger points are present.

CONTACTS AND LOCATIONS:
Overall Officials: Ziauddin University, Principal Investigator — Ziauddin
Locations (1):
- Ziauddin University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2017 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 354 diseases and injuries for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1789-1858. doi: 10.1016/S0140-6736(18)32279-7. Epub 2018 Nov 8. PMID 30496104
- [Background] Herekar AA, Ahmad A, Uqaili UL, Ahmed B, Effendi J, Alvi SZ, Shahab MA, Javed U, Herekar AD, Khanani R, Steiner TJ. Primary headache disorders in the adult general population of Pakistan - a cross sectional nationwide prevalence survey. J Headache Pain. 2017 Dec;18(1):28. doi: 10.1186/s10194-017-0734-1. Epub 2017 Feb 23. PMID 28229320
- [Background] Alonso-Blanco C, de-la-Llave-Rincon AI, Fernandez-de-las-Penas C. Muscle trigger point therapy in tension-type headache. Expert Rev Neurother. 2012 Mar;12(3):315-22. doi: 10.1586/ern.11.138. PMID 22364330
- [Background] Jensen RH. Tension-Type Headache - The Normal and Most Prevalent Headache. Headache. 2018 Feb;58(2):339-345. doi: 10.1111/head.13067. Epub 2017 Mar 13. PMID 28295304
- [Background] GBD 2015 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 310 diseases and injuries, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1545-1602. doi: 10.1016/S0140-6736(16)31678-6. PMID 27733282
- [Background] Kamali F, Mohamadi M, Fakheri L, Mohammadnejad F. Dry needling versus friction massage to treat tension type headache: A randomized clinical trial. J Bodyw Mov Ther. 2019 Jan;23(1):89-93. doi: 10.1016/j.jbmt.2018.01.009. Epub 2018 Jan 31. PMID 30691768
- [Background] Pourahmadi M, Mohseni-Bandpei MA, Keshtkar A, Koes BW, Fernandez-de-Las-Penas C, Dommerholt J, Bahramian M. Effectiveness of dry needling for improving pain and disability in adults with tension-type, cervicogenic, or migraine headaches: protocol for a systematic review. Chiropr Man Therap. 2019 Sep 26;27:43. doi: 10.1186/s12998-019-0266-7. eCollection 2019. PMID 31572570
- [Background] Shields G, Smith JM. Remedial Massage Therapy Interventions Including and Excluding Sternocleidomastoid, Scalene, Temporalis, and Masseter Muscles for Chronic Tension Type Headaches: a Case Series. Int J Ther Massage Bodywork. 2020 Feb 26;13(1):22-31. eCollection 2020 Mar. PMID 32133042
- [Background] Moraska AF, Stenerson L, Butryn N, Krutsch JP, Schmiege SJ, Mann JD. Myofascial trigger point-focused head and neck massage for recurrent tension-type headache: a randomized, placebo-controlled clinical trial. Clin J Pain. 2015 Feb;31(2):159-68. doi: 10.1097/AJP.0000000000000091. PMID 25329141
- [Background] Gildir S, Tuzun EH, Eroglu G, Eker L. A randomized trial of trigger point dry needling versus sham needling for chronic tension-type headache. Medicine (Baltimore). 2019 Feb;98(8):e14520. doi: 10.1097/MD.0000000000014520. PMID 30813155
- [Background] Munoz-Ceron J, Marin-Careaga V, Pena L, Mutis J, Ortiz G. Headache at the emergency room: Etiologies, diagnostic usefulness of the ICHD 3 criteria, red and green flags. PLoS One. 2019 Jan 7;14(1):e0208728. doi: 10.1371/journal.pone.0208728. eCollection 2019. PMID 30615622
- [Background] Overas CK, Myhrvold BL, Rosok G, Magnesen E. Musculoskeletal diagnostic ultrasound imaging for thickness measurement of four principal muscles of the cervical spine -a reliability and agreement study. Chiropr Man Therap. 2017 Jan 4;25:2. doi: 10.1186/s12998-016-0132-9. eCollection 2017. PMID 28070269
- [Background] Young IA, Dunning J, Butts R, Cleland JA, Fernandez-de-Las-Penas C. Psychometric properties of the Numeric Pain Rating Scale and Neck Disability Index in patients with cervicogenic headache. Cephalalgia. 2019 Jan;39(1):44-51. doi: 10.1177/0333102418772584. Epub 2018 Apr 19. PMID 29673262